CLINICAL TRIAL: NCT02810288
Title: A Survey of Airway Management Practice Patterns in Paediatric Anaesthesia by Anaesthesiologists in Different European Hospitals
Brief Title: Airway Management Practice Patterns in Paediatric Anaesthesia: A Survey
Acronym: SUR-AMPA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Thekla Niebel, MD PhD, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: AR-01-SUR-AMPA
Record Dates: First submitted 2016-06-14; First posted 2016-06-22 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Paediatric Airway Management
Keywords: Airway anatomy; difficult intubation; congenital syndromes

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Expert: Anaesthesiologist with large paediatric daily practice. All participant voluntarily response all items in the questionnaire database.
  Interventions: Behavioral: Voluntarily response all items in the questionnaire.
- Non-experts: Anaesthesiologist with little paediatric daily practice. All participant voluntarily response all items in the questionnaire database.
  Interventions: Behavioral: Voluntarily response all items in the questionnaire.

INTERVENTIONS:
Behavioral: Voluntarily response all items in the questionnaire. — The study type is a cross-sectional study, by means of electronic self-administered survey as online questionnaire sent by e-mail.
  The questionnaire for the survey was developed with reference to previously published guidelines on the design of questionnaire surveys. The content validity of the questionnaire was verified by review of clinicians not participating into the project and by a statistician.

SUMMARY:
Respiratory adverse events continue to be the leading reason for perioperative critical events in children. It is crucial for the anaesthesiologist to anticipate, recognize and treat these respiratory adverse events. Respiratory adverse events are one of the major causes of morbidity and mortality during paediatric anaesthesia. To avoid trouble, one must be prepared for trouble: if a difficult airway is very likely, anaesthesia should be administered by experienced anaesthesiologists and should only be performed in a protected well-equipped area where the personnel adequately trained.

This survey focuses on assessment and management of paediatric airway and highlights the unique challenges encountered in children.

DETAILED DESCRIPTION:
Airway management is one of the key areas of paediatric anaesthesia practice. The paediatric patients have significant anatomical and physiological differences compared with adults, which impact on the techniques and tools that the anaesthesiologist might choose to provide safe and effective control of the airway. Furthermore, there are a number of pathological processes, typically seen in the paediatric population, which present unique anatomical or functional difficulties in airway management. The presence of one of these syndromes or conditions can predict a "difficult airway".

Respiratory adverse events continue to be the leading reason for perioperative critical events in children. New developments in airway management in paediatric patients can only improve perioperative outcome if anaesthesiologists who are fully acquainted with these fundamental aspects of paediatric anaesthesia care for these children.

This survey was taken out within members of the Community of European Anaesthesiologists, to describe and explore current patterns of their airway management in paediatric anaesthesia.

The purpose of the study was to see whether there are more uniform practice patterns among anaesthesiologist with paediatric experience than those without paediatric experience.

Secondarily, the survey also explored anaesthetists'' knowledge about the risks of respiratory adverse events and, and about national organizations' recommendations.

Therefore, this survey highlighted some of the important anatomical and physiological differences and their implication in daily anaesthesiological practice.

ELIGIBILITY:
Inclusion Criteria:

* Anaesthesiologists currently working in the operating rooms.

Exclusion Criteria:

* unwilling to join the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Volunteers among the anaesthesiological community of 5 different European countries. All participant voluntarily response all items in the questionnaire database.
  A representative anaesthesiologist for each of the target Countries will be asked to participate and to invite at least one other hospital. All anaesthesiologists within each selected hospital will be asked to participate in the survey.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of anaesthesiologist with paediatric experience using intravenous induction compared to those without paediatric experience. | A time of survey; generally less than 20 minutes
  The primary objective will be to compare anaesthesiologists with and without paediatric experience in terms of proportion of anaesthesiologists adopting "standard" practice.

SECONDARY OUTCOMES:
Proportion of anaesthesiologist with paediatric experience measuring cuff pressure with pressure manometer compared to those without paediatric experience. | A time of survey; generally less than 20 minutes
  The objective will be to compare anaesthesiologists with and without paediatric experience in terms of proportion of anaesthesiologists adopting "standard" practice.
Proportion of participants correctly identifying predictability of difficult airway in children. | A time of survey; generally less than 20 minutes
  To assess variables associated to adoption of standard practice, in particular: knowledge of the anatomical, physiological, and pathological features related to the airway.
Proportion of participants correctly answering questions about the use of (modified) rapid sequence induction in the paediatric population. | A time of survey; generally less than 20 minutes
  To compare anaesthesiologists with and without paediatric experience in terms of different practice patterns, and items explored by the questionnaire.
Proportion of anaesthesiologist correctly identifying national organisations difficult airway recommendations. | A time of survey; generally less than 20 minutes
  To informally compare practiced elicited within this study to existing guidelines and algorithms in paediatric anaesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Braschi, MD Prof, Study Chair — IRCCS Policlinico San Matteo
Locations (1):
- IRCCS Policlinico San Matteo, Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clergue F, Auroy Y, Pequignot F, Jougla E, Lienhart A, Laxenaire MC. French survey of anesthesia in 1996. Anesthesiology. 1999 Nov;91(5):1509-20. doi: 10.1097/00000542-199911000-00045. PMID 10551604
- [Background] Auroy Y, Ecoffey C, Messiah A, Rouvier B. Relationship between complications of pediatric anesthesia and volume of pediatric anesthetics. Anesth Analg. 1997 Jan;84(1):234-5. doi: 10.1097/00000539-199701000-00060. No abstract available. PMID 8989044
- [Background] Harless J, Ramaiah R, Bhananker SM. Pediatric airway management. Int J Crit Illn Inj Sci. 2014 Jan;4(1):65-70. doi: 10.4103/2229-5151.128015. PMID 24741500
- [Background] Von Ungern-Sternberg BS, Habre W. Pediatric anesthesia - potential risks and their assessment: part I. Paediatr Anaesth. 2007 Mar;17(3):206-15. doi: 10.1111/j.1460-9592.2006.02097.x. No abstract available. PMID 17263734
- [Background] Burns KE, Duffett M, Kho ME, Meade MO, Adhikari NK, Sinuff T, Cook DJ; ACCADEMY Group. A guide for the design and conduct of self-administered surveys of clinicians. CMAJ. 2008 Jul 29;179(3):245-52. doi: 10.1503/cmaj.080372. No abstract available. PMID 18663204
- [Background] van Gelder MM, Bretveld RW, Roeleveld N. Web-based questionnaires: the future in epidemiology? Am J Epidemiol. 2010 Dec 1;172(11):1292-8. doi: 10.1093/aje/kwq291. Epub 2010 Sep 29. PMID 20880962
- [Background] Kelley K, Clark B, Brown V, Sitzia J. Good practice in the conduct and reporting of survey research. Int J Qual Health Care. 2003 Jun;15(3):261-6. doi: 10.1093/intqhc/mzg031. PMID 12803354
- [Background] Tait AR, Voepel-Lewis T. Survey research: it's just a few questions, right? Paediatr Anaesth. 2015 Jul;25(7):656-62. doi: 10.1111/pan.12680. Epub 2015 Apr 30. PMID 25929546
- [Background] Hohne C, Haack M, Machotta A, Kaisers U. [Airway management in pediatric anesthesia]. Anaesthesist. 2006 Jul;55(7):809-19; quiz 820. doi: 10.1007/s00101-006-1045-0. German. PMID 16804684